CLINICAL TRIAL: NCT01684605
Title: A Randomized, Double-blind, Active Control, Single Dosing, Crossover Clinical Trial to Investigate the Pharmacokinetics of CKD-11101 and NESP After IV Administration in Health Male Volunteers
Brief Title: Pharmacokinetics Study of CKD-11101 and NESP After IV Administration in Health Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 136HPS12D
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Anemia
Keywords: CKD-11101; NESP; Darbepoetin alfa; Anemia; intravenous; Pharmacokinetics; Phase 1
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NESP 60μg (Active Comparator): Prefilled syringe filled with Darbepoetin alfa 60μg
  Interventions: Drug: NESP 60μg
- CKD-11101 60μg (Experimental): Prefilled syringe filled with Darbepoetin alfa 60μg
  Interventions: Drug: CKD-11101 60μg

INTERVENTIONS:
Drug: NESP 60μg — Administrated NESP 60μg once intravenously
  Arms: NESP 60μg
Drug: CKD-11101 60μg — Administrated CKD-11101 60μg once intravenously
  Arms: CKD-11101 60μg

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of CKD-11101 and NESP after IV administration in health male volunteers

DETAILED DESCRIPTION:
Healthy volunteers are administrated CKD-11101 60μg and NESP 60μg once intravenously. (crossover) Every time before and after taking each medication, PK parameters and safety of CKD-11101 60μg and NESP 60μg are performed using a blood sample and conducting some tests(Laboratory test, V/S and Physical Examination, etc) respectively.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form prior to study participation.
* A healthy male volunteer between 20 and 55 years old.
* Body weight between 55kg and 90kg, BMI between 18 and 27.
* Appropriate subject for the study judging from investigator(physical examination, laboratory test, interview, etc.)

Exclusion Criteria:

* Have the medical history of allergic diseases including hypersensitivity against drug or clinically significant allergic diseases
* Clinically significant hepatic, renal, respiratory system, endocrine system, nervous system, immune system, hematologic, psychiatric, circulatory system, tumor or have history of tumor
* Have abnormal laboratory result.

  * Hemoglobin < 12g/dL or > 17g/dL
  * Vitamin B12 < 200pg/mL
  * Ferritin < 21.8ng/mL
  * Transferrin < 190mg/dL
  * Reticulocyte over the normal limit
  * Positive for the Triage TOX drug on urine (cocaine, amphetamines, barbiturates, opiates, benzodiazepine, cannabinoids)
  * Positive for HIV antibody, HBsAg, HCV antibody test
* A heavy smoker (cigarette > 10 cigarettes per day)
* Administer EPO, darbepoetin, immunoglobulin or IV iron within 3 months prior to the first IP administration
* Have hypersensitivity reactions history for EPO, darbepoetin, excipient of IP or iron tablets
* sit SBP < 90mmHg or sit SBP > 140mmHg or sit DBP < 55mmHg or sit DBP > 90mmHg or Pulse rate > 100 per/min
* History of hemoglobinopathy or inflammatory disease or drug abuse within 6 months before screening
* Subject takes ethical drug or herbal medicine within 14 days, OTC or vitamin supplements within 7 days before the first IP administration
* Participated in the other clinical trials and administrated IP within 8 weeks prior to the first IP administration
* A heavy alcohol consumer (alcohol > 21 units/week) or cannot stop drinking
* Bleed or donate blood (> 400mL) within 8 weeks before the first IP administration
* Participated in this clinical trials and administrated IP
* Have a diet within 2 days before the first IP administration or cannot stop having

  * food containing grapefruit
  * food containing caffeine
* Disagree to avoid getting pregnant during clinical trial
* An impossible one who participates in clinical trial by investigator's decision including laboratory test result, other reason

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2012-10-12 (Actual); Primary Completion 2012-11-13 (Actual); Study Completion 2013-01-03 (Actual)

PRIMARY OUTCOMES:
Assess AUClast of darbepoetin alfa | Pre-dose, 0.25h, 0.5h, 0.75h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 72h, 96h, 120h, 168h, 264h
Assess Cmax of darbepoetin alfa | Pre-dose, 0.25h, 0.5h, 0.75h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 72h, 96h, 120h, 168h, 264h

SECONDARY OUTCOMES:
Assess AUCinf of darbepoetin alfa | Pre-dose, 0.25h, 0.5h, 0.75h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 72h, 96h, 120h, 168h, 264h
Assess Tmax of darbepoetin alfa | Pre-dose, 0.25h, 0.5h, 0.75h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 72h, 96h, 120h, 168h, 264h
Assess t1/2 of darbepoetin alfa | Pre-dose, 0.25h, 0.5h, 0.75h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 72h, 96h, 120h, 168h, 264h
Assess CL of darbepoetin alfa | Pre-dose, 0.25h, 0.5h, 0.75h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 72h, 96h, 120h, 168h, 264h

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Sang Yu, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea